CLINICAL TRIAL: NCT00870987
Title: Clinical Trial on Safety, Immunogenicity, and Efficacy of a Prime Boost Regimen of DNA- and Adenovirus-vectored Malaria Vaccines Encoding Plasmodium Falciparum Circumsporozoite Protein and Apical Membrane Antigen 1 in Healthy Malaria-Naïve Adults in the US
Brief Title: Clinical Trial for Malaria Vaccines to Test for Safety, Immune Response and Protection Against Malaria
Acronym: DNA-Ad
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WRAIR 1550; HRPO #A-15350; NMRC.2009.0004
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Malaria
Keywords: Malaria; Vaccine
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): DNA vaccine prime Given at 0, 4, and 8 weeks
  Interventions: Biological: DNA vaccine prime
- 2 (Experimental): adenovirus type 5 vaccine boost Given at 24 weeks
  Interventions: Biological: adenovirus type 5 vaccine boost

INTERVENTIONS:
Biological: DNA vaccine prime — 2 mg total dose (1 mg per construct in a volume of 1 mL)
  Arms: 1
Biological: adenovirus type 5 vaccine boost — 2 x 1010 particle units (pu) (1 x 1010 pu per each of 2 constructs including CSP and AMA1 respectively)
  Arms: 2

SUMMARY:
The purpose of this study is to test the safety and effectiveness of a new malaria vaccine, the DNA-Ad vaccine. The study is specifically looking at a vaccine regimen against Plasmodium falciparum, the most deadly form of malaria.

DETAILED DESCRIPTION:
The goal of this study is to evaluate if the DNA-Ad vaccine that targets both the liver and blood stages of the malaria life cycle is safe and protective, in hopes to develop a vaccine to prevent infection and/or lessen the severity of disease caused by the P. falciparum malaria parasite. More specifically, this DNA-Ad vaccine contains a liver stage antigen (circumsporozoite protein) and an antigen (apical membrane antigen 1) that is present in both the liver and blood stages designed to prevent infection by killing the majority of developing parasites in the liver and to prevent severe disease and death should break-through blood stage infections occur.

This study is an open-label, Phase 1/2a study designed to assess the safety, immunogenicity, and efficacy of a DNA-Ad vaccine in healthy adults who are Ad5 seropositive or seronegative. The vaccinated study group will consist of up to 20 healthy, malaria-naïve adults aged 18 to 50 years, who have been previously screened to meet inclusion and exclusion criteria and will receive three priming doses of the DNA vaccine and a single dose of the boosting component, an adenovirus-vectored vaccine to be given 4 months after the last dose of DNA. Follow up visits will occur after each immunization. The control group will consist of six non-immunized subjects that will participate in a challenge to assure that vaccinated subjects were indeed exposed to P. falciparum. Subjects in both the immunized and control cohorts will receive malaria challenge. Subjects will be assessed for development of parasitemia by daily blood smears and will be closely observed in hotel after the challenge. Subjects will then be followed periodically and have the final in-person visit twelve weeks after the challenge, followed by annual contact by phone, email, or mailings up to five years after the first dose of immunization per FDA recommendation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18 to 50 years of age (inclusive)
* Women who are not pregnant by a current negative pregnancy test or of non-childbearing potential
* Willing to use an FDA approved birth control method including condoms, birth control pills, sterility surgery, or intrauterine devices among others, from time of enrollment until 6 months after the end of the active phase of the study
* Able to provide free and willing written informed consent to participate
* Score at least 80% correct on a 10 question Assessment of Understanding
* No plans to travel to a malaria endemic area during the course of the study
* Free of significant health problems as established by medical history and clinical examination completed prior to the study
* Available to participate and reachable for duration of study (up to five years)
* Only subjects with no or low cardiac risk factors according to the Gaziano study [53] and a normal EKG will be included in the study

Exclusion Criteria:

* Pregnant (positive HCG) or nursing at screening or plans to become pregnant or nurse from the time of enrollment until 6 months after sporozoite challenge
* Any past history of malaria
* History of receipt of malaria vaccine
* Plans to travel to malarious areas during the study period
* Use of any investigational or non-registered drug or vaccine within 30 days prior to enrollment
* Seropositive for HIV, hepatitis C virus (antibodies to HIV and HCV), and/or HBsAg
* Subjects in the immunized group who engage in high-risk behaviors for acquiring HIV
* Allergy to antimalarials or significant (e.g. systemic) hypersensitivity reactions to mosquito bites (local hypersensitivity reactions at the site of a mosquito bite are not an exclusion criterion)
* History of psoriasis (given its interaction with chloroquine)
* Use or planned use of any drugs with significant anti-malarial activity, such as doxycycline, clindamycin, azithromycin, or trimethoprim/sulfamethoxazole among others during the study period (subjects can withhold the use of these medications during the study period if approved by their primary care physicians, at the minimum starting from four weeks before vaccine administration until four weeks after becoming parasitemic) Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection and history of splenectomy
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying drugs within six months of challenge
* A family history of congenital or hereditary immunodeficiency
* Chronic or active neurologic disease including seizure disorder
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by medical history, physical examination, or abnormal baseline laboratory screening tests.
* Abnormal baseline EKG obtained at screening
* Acute disease at the time of enrollment
* Hepatomegaly, right upper quadrant abdominal pain or tenderness: noted by physical exam during the screening process.
* Administration of immunoglobulins and/or any blood products within the three months preceding immunization during the study period
* Use of kanamycin or related antibiotics
* Suspected or known current alcohol abuse/drug abuse as obtained by history and physical examination
* Inability to make follow-up visits
* Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 5 years
  The vaccine will be considered safe and well-tolerated if there are no severe or serious adverse events (AE) related to vaccine administration or if any severe events are relatively benign (e.g.
  erythema meeting criteria for severe due to its dimensions but not significantly affecting the activities of daily living for the subject) or brief in duration (e.g. less than 48 hours). The AEs will be assessed according to the method below.
  1. Occurrence, severity, and duration of any solicited symptoms starting on the day of immunization through day 7 after each immunization
  2. Occurrence of any unsolicited symptoms, abnormal physical findings, and laboratory values starting from the day of immunization through day 28 after each immunization
  3. Occurrence of any serious adverse events, as defined in 21 CFR 312.32, during the five-year study period

SECONDARY OUTCOMES:
Number of sterile or partial protections | 28 days after malaria challenge
  The DNA-Ad vaccine is considered efficacious if it offers any degree of sterile or partial protection that reaches statistical significance (p<0.05). The vaccine efficacy will be determined by two parameters: 1) sterile protection for 28 days after challenge, 2) partial protection as determined by delay to parasitemia by smears and PCR.
Number of humoral immunity expressions | 28 days after malaria challenge
  The DNA-Ad vaccine is considered to confer humoral immunity if the increase of antibody response for CSP or AMA1 by ELISA post immunization is statistically significant (p<0.05) compared to the levels before immunization.
Number of cellular immunity expressions | 28 days after malaria challenge
  The DNA-Ad vaccine is considered to confer cellular immunity if a positive ELISpot response is detected after immunization

CONTACTS AND LOCATIONS:
Overall Officials: Judith Epstein, MD, Principal Investigator — US Military Vaccine Program, NMRC PI, Naval Officer
Locations (1):
- Clinical Trials Center, WRAIR, Silver Spring, Maryland, United States

REFERENCES:
- [Derived] Sedegah M, Peters B, Hollingdale MR, Ganeshan HD, Huang J, Farooq F, Belmonte MN, Belmonte AD, Limbach KJ, Diggs C, Soisson L, Chuang I, Villasante ED. Vaccine Strain-Specificity of Protective HLA-Restricted Class 1 P. falciparum Epitopes. PLoS One. 2016 Oct 3;11(10):e0163026. doi: 10.1371/journal.pone.0163026. eCollection 2016. PMID 27695088
- [Derived] Aguiar JC, Bolton J, Wanga J, Sacci JB, Iriko H, Mazeika JK, Han ET, Limbach K, Patterson NB, Sedegah M, Cruz AM, Tsuboi T, Hoffman SL, Carucci D, Hollingdale MR, Villasante ED, Richie TL. Discovery of Novel Plasmodium falciparum Pre-Erythrocytic Antigens for Vaccine Development. PLoS One. 2015 Aug 20;10(8):e0136109. doi: 10.1371/journal.pone.0136109. eCollection 2015. PMID 26292257
- [Derived] Sedegah M, Hollingdale MR, Farooq F, Ganeshan H, Belmonte M, Huang J, Abot E, Limbach K, Chuang I, Tamminga C, Epstein JE, Villasante E. Controlled Human Malaria Infection (CHMI) differentially affects cell-mediated and antibody responses to CSP and AMA1 induced by adenovirus vaccines with and without DNA-priming. Hum Vaccin Immunother. 2015;11(11):2705-15. doi: 10.1080/21645515.2015.1019186. Epub 2015 Aug 20. PMID 26292027
- [Derived] Sedegah M, Hollingdale MR, Farooq F, Ganeshan H, Belmonte M, Kim Y, Peters B, Sette A, Huang J, McGrath S, Abot E, Limbach K, Shi M, Soisson L, Diggs C, Chuang I, Tamminga C, Epstein JE, Villasante E, Richie TL. Sterile immunity to malaria after DNA prime/adenovirus boost immunization is associated with effector memory CD8+T cells targeting AMA1 class I epitopes. PLoS One. 2014 Sep 11;9(9):e106241. doi: 10.1371/journal.pone.0106241. eCollection 2014. PMID 25211344
- [Derived] Tamminga C, Sedegah M, Maiolatesi S, Fedders C, Reyes S, Reyes A, Vasquez C, Alcorta Y, Chuang I, Spring M, Kavanaugh M, Ganeshan H, Huang J, Belmonte M, Abot E, Belmonte A, Banania J, Farooq F, Murphy J, Komisar J, Richie NO, Bennett J, Limbach K, Patterson NB, Bruder JT, Shi M, Miller E, Dutta S, Diggs C, Soisson LA, Hollingdale MR, Epstein JE, Richie TL. Human adenovirus 5-vectored Plasmodium falciparum NMRC-M3V-Ad-PfCA vaccine encoding CSP and AMA1 is safe, well-tolerated and immunogenic but does not protect against controlled human malaria infection. Hum Vaccin Immunother. 2013 Oct;9(10):2165-77. doi: 10.4161/hv.24941. Epub 2013 Jun 4. PMID 23899517
- [Derived] Chuang I, Sedegah M, Cicatelli S, Spring M, Polhemus M, Tamminga C, Patterson N, Guerrero M, Bennett JW, McGrath S, Ganeshan H, Belmonte M, Farooq F, Abot E, Banania JG, Huang J, Newcomer R, Rein L, Litilit D, Richie NO, Wood C, Murphy J, Sauerwein R, Hermsen CC, McCoy AJ, Kamau E, Cummings J, Komisar J, Sutamihardja A, Shi M, Epstein JE, Maiolatesi S, Tosh D, Limbach K, Angov E, Bergmann-Leitner E, Bruder JT, Doolan DL, King CR, Carucci D, Dutta S, Soisson L, Diggs C, Hollingdale MR, Ockenhouse CF, Richie TL. DNA prime/Adenovirus boost malaria vaccine encoding P. falciparum CSP and AMA1 induces sterile protection associated with cell-mediated immunity. PLoS One. 2013;8(2):e55571. doi: 10.1371/journal.pone.0055571. Epub 2013 Feb 14. PMID 23457473